CLINICAL TRIAL: NCT03641053
Title: Comparison of Honey and Povidone-iodine in Wound Healing on Acute Laceration Wounds: A Randomized Controlled Trial Study
Brief Title: Honey Versus Povidone-iodine on Laceration Wounds
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: S.K. Lerik General Hospital (Other)
Responsible Party: Principal Investigator, Kevin Leonard Suryadinata, Kevin Leonard Suryadinata, MD. Principal Investigator and General Practitioner of S.K. Lerik General Hospital, S.K. Lerik General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKL001
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Laceration Face; Wound Heal; Wounds and Injuries; Laceration Arm; Laceration of Leg
Keywords: honey; povidone-iodine; randomized control trial; wound healing
MeSH Terms: conditions — Wounds and Injuries | interventions — Honey; Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: A three-arm parallel assignment where one group receives honey, the second group receives povidone-iodine, and the third group receives paraffin gauze as wound dressing.
Who Masked: Participant
Masking Description: Participants do not know which intervention substance they have been assigned to
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Honey (Experimental): 0.05 cc of honey (Madu Nusantara®) per 1 cm of laceration, given every predetermined wound care schedule
  Interventions: Other: Honey
- Povidone-iodine (Active Comparator): 0.05 cc of povidone-iodine per 1 cm of laceration, given every predetermined wound care schedule
  Interventions: Other: Povidone-iodine
- Paraffin gauze (Active Comparator): 1 layer of paraffin gauze, given every predetermined wound care schedule
  Interventions: Other: Paraffin gauze

INTERVENTIONS:
Other: Honey — Substance is given topically after the wound has been sutured
  Other Names: Madu Nusantara®
  Arms: Honey
Other: Povidone-iodine — Substance is given topically after the wound has been sutured
  Other Names: OneMed® povidone-iodine 10%
  Arms: Povidone-iodine
Other: Paraffin gauze — Substance is given topically after the wound has been sutured
  Other Names: Cuticell® Classic Paraffin Gauze
  Arms: Paraffin gauze

SUMMARY:
This study evaluates healing time in usage of honey and povidone-iodine over paraffin gauze as dressings in the treatment of acute laceration wounds. In Indonesia, especially in rural area, where most of the resources is limited and modern dressings are expensive and hard-to-find. The investigators tried to find an alternative which was easier to find and could act as a substitute of modern wound dressing.

The hypothesis of this study is honey and povidone-iodine could be a good substitute (or equal to) to paraffin gauze on acute laceration wounds.

Honey is chosen because of its versatility and already well-known to be used as a chronic wound dressing. Povidone-iodine was chosen as another alternative because it is still one of the most used substance in rural area as a wound dressing, but there is not enough study to support the usage of this substance. Paraffin gauze was chosen as a representative of modern wound dressing because it fulfilled the standard of wound dressing on acute wound, which is non-adherent and also moist.

DETAILED DESCRIPTION:
The investigator's team consists of five members, each have their own specific tasks and divided by two groups, which are ER group (first time encounter, informed consent, and intervention) and polyclinic group (routine wound care). All of the data are primary data. Data registry were taken by the team without involving any other party. Any intervention done to the participants were also done only by the team(suturing, wound care). Appointment for routine wound care was also made by contacting the participant through their cellphone numbers which were collected when they come to the ER.

The data of each of the participant was registered on a form which was pre-made by the investigators. It recorded the identity of the patient, history taking, physical examination, and also to record more detailed information about our intervention, such as the amount of stitches and how many and what kind of resources that have been spent on the participant.

Every sample will be categorized into 3 randomized groups of intervention; honey, povidone-iodine, and paraffin gauze, which will also be categorized by location of their wound; face and neck, upper extremity, and lower extremity. Participants on each intervention group are distributed evenly using stratified block randomization. Photos of the wound will be taken before and after the wound is cleaned, and after the wound has been sutured. Every patient will be asked to attend a predetermined schedule for wound care assessment. The wound will be evaluated by photos before and after the wound is cleaned, debrided, or have its sutures removed. Parameter of evaluation will be duration of wound healing per anatomical region, infection, cleanliness of wound, odor, exudate level, pain, itch, and total cost of wound care.

Every paper consists of participants' data that were collected on colored maps based on the intervention group (red: povidone-iodine, yellow: honey, blue: paraffin). At the end of the study, three of the team's members converted the data to be analyzed using Microsoft Excel and SPSS.

The investigators prepared beforehand the Standard Operational Procedures regarding any possibilities of adverse events, such as lidocaine toxicity and honey hypersensitivity and were already approved by the hospital's committee.

The investigators determined the target of the sample size with the total sample of 36 participants, distributed evenly based on intervention groups and wounds' location using stratified block randomization

ELIGIBILITY:
Inclusion Criteria:

Every patient that admits to the emergency department with:

* An acute open traumatic wound
* Agrees to a voluntary agreement for informed consent
* To be treated in an outpatient setting

Exclusion Criteria:

Human factor:

* Patient under the age of 10 and over 60 years old
* Systemic conditions (diabetes mellitus, hypertension, liver' kidney disease)
* Signs of infection
* Consuming steroids and / or antibiotics
* History of keloid
* History of drug and / or alcohol abuse
* Under treatment for chemotherapy or immunocompromised
* Pregnant
* History of allergy towards amoxicillin and / or ibuprofen

Wound factor:

* Acute Open Traumatic Wound that has occured after than 12 hours of admittance to the emergency department
* Open fracture
* Suspicion of contamination from the mechanism of attaining the wound (human or animal bite, body fluids such as faeces, saliva, urine, sperm, or vaginal secretion)
* Penetration trauma (stab wound, gunshot wound, or a joint-affected wound)
* Signs of wound infection
* More than one wound in the same anatomical region
* Possess a chronic wound caused by underlying disease other than trauma
* Wound with exposed tendon and/ or bone
* Wound length dimension no less than 1 cm and no more than 10 cm.
* Hypersensitivity to honey
* Does not attend to scheduled wound care assesment control
* Sample's wish to not be involved anymore with the research at any phase

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Wound healing time | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured by days, when was all of the sutures completely removed and the wound is completely approximated. We followed the guideline from American Academy of Family Physicians for timing for suture removal, so we will not remove the suture before the recommended time

SECONDARY OUTCOMES:
Infection | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured using the infection signs from Delphi Criteria
Pain level | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  measured using Numeral Rating Scale from 0-10, asked from the onset of the wound and every routine wound care
Itchiness | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured using Numeral Rating Scale from 0-10, asked from the onset of the wound and every routine wound care
Odor | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured using Verbal Rating Scale, consists of 4 level of odor (no odor, slight odor, medium odor, strong odor), asked from the onset of the wound and every routine wound care
Exudate | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured in grams, using digital scale with the precision of 3 digits. We measured the gauze which will be used and the one which is already on top the wound, from the onset of the wound and every routine wound care
Cleanliness | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured using images taken from the whole photographs of the wound. This parameter was measured using "less clean", "cleaner", "unchanged cleanliness". statistically using Cohen's kappa score to reach the agreement of the evaluation of this parameter
Cost | 28 days/4 weeks; day 0 is the day of the event. The participants was chosen very carefully by our strict eligibility criteria, so the investigators expect that the wound will heal on acute period
  Measured by counting the cost of every material used for the participant

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Suryadinata, MD, Principal Investigator
Locations (1):
- S.K. Lerik General Hospital, Kupang, East Nusa Tenggara, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fife CE, Carter MJ. Wound Care Outcomes and Associated Cost Among Patients Treated in US Outpatient Wound Centers: Data From the US Wound Registry. Wounds. 2012 Jan;24(1):10-7. PMID 25875947
- [Background] Sood A, Granick MS, Tomaselli NL. Wound Dressings and Comparative Effectiveness Data. Adv Wound Care (New Rochelle). 2014 Aug 1;3(8):511-529. doi: 10.1089/wound.2012.0401. PMID 25126472
- [Background] Dhivya S, Padma VV, Santhini E. Wound dressings - a review. Biomedicine (Taipei). 2015 Dec;5(4):22. doi: 10.7603/s40681-015-0022-9. Epub 2015 Nov 28. PMID 26615539
- [Background] Indonesia | Data. Indonesia [Internet]. 2017 [updated 2017; cited 2017 Jun 18]. Available from: http://data.worldbank.org/country/indonesia.
- [Background] Trihono. Riset Kesehatan Dasar: Riskesdas 2013. Jakarta: Badan Penelitian dan Pengembangan Kesehatan Kementerian Kesehatan RI.
- [Background] Produk Domestik Bruto - Analisis PDB Per Kapita Indonesia | Indonesia Investments. Produk Domestik Bruto Indonesia [Internet]. 2017 [updated 2017 Feb 6; cited 2017 Jun 18]. Available from: https://www.indonesia-investments.com/id/keuangan/angka-ekonomi-makro/produk-domestik-bruto-indonesia/item253.
- [Background] Badan Pusat Statistik. Upah Minimum Regional/Provinsi (UMR/UMP) dan rata-rata Nasional per tahun (Dalam Rupiah), 1997-2016 [Internet]. Jakarta: Badan Pusat Statistik; 2016 [updated 2016; cited 2017 Jun 18]. Available from: https://www.bps.go.id/linkTableDinamis/view/id/917
- [Background] Moeloek NF. Peraturan Menteri Kesehatan Republik Indonesia Nomor 4 Tahun 2017 Tentang Perubahan Kedua Atas Peraturan Menteri Kesehatan Nomor 52 Tahun 2016 Tentang Standar Tarif Pelayanan Kesehatan Dalam Penyelenggaraan Program Jaminan Kesehatan. Jakarta: Menteri Kesehatan Republik Indonesia; 2017. pg. 6.
- [Background] Hemani ML, Lepor H. Skin preparation for the prevention of surgical site infection: which agent is best? Rev Urol. 2009 Fall;11(4):190-5. PMID 20111631
- [Background] Angel DE, Morey P, Storer JG, Mwipatayi BP. The great debate over iodine in wound care continues: a review of the literature. Wound Pract Res. 2008;16(1):6-21.
- [Background] Jull AB, Walker N, Deshpande S. Honey as a topical treatment for wounds. Cochrane Database Syst Rev. 2013 Feb 28;(2):CD005083. doi: 10.1002/14651858.CD005083.pub3. PMID 23450557
- [Background] Saikaly SK, Khachemoune A. Honey and Wound Healing: An Update. Am J Clin Dermatol. 2017 Apr;18(2):237-251. doi: 10.1007/s40257-016-0247-8. PMID 28063093
- [Background] Nevas M, Lindstrom M, Horman A, Keto-Timonen R, Korkeala H. Contamination routes of Clostridium botulinum in the honey production environment. Environ Microbiol. 2006 Jun;8(6):1085-94. doi: 10.1111/j.1462-2920.2006.001000.x. PMID 16689729
- [Background] Shukrimi A, Sulaiman AR, Halim AY, Azril A. A comparative study between honey and povidone iodine as dressing solution for Wagner type II diabetic foot ulcers. Med J Malaysia. 2008 Mar;63(1):44-6. PMID 18935732
- [Background] Gulati S, Qureshi A, Srivastava A, Kataria K, Kumar P, Ji AB. A Prospective Randomized Study to Compare the Effectiveness of Honey Dressing vs. Povidone Iodine Dressing in Chronic Wound Healing. Indian J Surg. 2014 Jun;76(3):193-8. doi: 10.1007/s12262-012-0682-6. Epub 2012 Jul 12. PMID 25177115
- [Background] Li J, Chen J, Kirsner R. Pathophysiology of acute wound healing. Clin Dermatol. 2007 Jan-Feb;25(1):9-18. doi: 10.1016/j.clindermatol.2006.09.007. PMID 17276196
- [Background] Thorne CHM, Gurtner GC, Chung K, Gosain A Mehrara B, Rubin P, Spear SL Grabb and Smith's Plastic Surgery. 7th ed.. Lippincott Williams & Wilkins, Philadelphia, USA. Pg. 14-17.
- [Background] Siddiqui AR, Bernstein JM. Chronic wound infection: facts and controversies. Clin Dermatol. 2010 Sep-Oct;28(5):519-26. doi: 10.1016/j.clindermatol.2010.03.009. PMID 20797512
- [Background] Kumar V, Cotran RS, Robbin ST. Robbins basic Pathology. 7th ed. Philadelphia, 2003, Saunders.
- [Background] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Background] Troxler M, Vowden K, Vowden P. 2006. Integrating Adjunctive Therapy into Practice: The Importance of Recofnising 'Hard-to-Heal' Wounds.
- [Background] Lazarus GS, Cooper DM, Knighton DR, Percoraro RE, Rodeheaver G, Robson MC. Definitions and guidelines for assessment of wounds and evaluation of healing. Wound Repair Regen. 1994 Jul;2(3):165-70. doi: 10.1046/j.1524-475X.1994.20305.x. PMID 17156107
- [Background] Fonseca JA et al. Medscape Education. Burn Wound Infections. [Online]. Updated May 25, 2016. Available at http://emedicine.medscape.com/article/213595-overview. Accessed June 16, 2017.
- [Background] Nicks BA, Ayello EA, Woo K, Nitzki-George D, Sibbald RG. Acute wound management: revisiting the approach to assessment, irrigation, and closure considerations. Int J Emerg Med. 2010 Aug 27;3(4):399-407. doi: 10.1007/s12245-010-0217-5. PMID 21373312
- [Background] Yaghoobi R, Kazerouni A, Kazerouni O. Evidence for Clinical Use of Honey in Wound Healing as an Anti-bacterial, Anti-inflammatory Anti-oxidant and Anti-viral Agent: A Review. Jundishapur J Nat Pharm Prod. 2013 Aug;8(3):100-4. doi: 10.17795/jjnpp-9487. Epub 2013 Jul 17. PMID 24624197
- [Background] Kaufman T, Eichenlaub EH, Angel MF, Levin M, Futrell JW. Topical acidification promotes healing of experimental deep partial thickness skin burns: a randomized double-blind preliminary study. Burns Incl Therm Inj. 1985 Dec;12(2):84-90. doi: 10.1016/0305-4179(85)90032-4. PMID 4092157
- [Background] Greener B, Hughes AA, Bannister NP, Douglass J. Proteases and pH in chronic wounds. J Wound Care. 2005 Feb;14(2):59-61. doi: 10.12968/jowc.2005.14.2.26739. No abstract available. PMID 15739652
- [Background] Biswas A, Bharara M, Hurst C, Gruessner R, Armstrong D, Rilo H. Use of sugar on the healing of diabetic ulcers: a review. J Diabetes Sci Technol. 2010 Sep 1;4(5):1139-45. doi: 10.1177/193229681000400512. PMID 20920433
- [Background] Molan P, Rhodes T. Honey: A Biologic Wound Dressing. Wounds. 2015 Jun;27(6):141-51. PMID 26061489
- [Background] Portenoy RK, Tanner RM. Pain Management: Theory and Practice. Oxford: Oxford University Press; 1996.
- [Background] Bijur PE, Latimer CT, Gallagher EJ. Validation of a verbally administered numerical rating scale of acute pain for use in the emergency department. Acad Emerg Med. 2003 Apr;10(4):390-2. doi: 10.1111/j.1553-2712.2003.tb01355.x. PMID 12670856
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03641053/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT03641053/ICF_001.pdf